CLINICAL TRIAL: NCT04117373
Title: Characterizing Trends in Mohs Micrographic Surgery and Complex Reconstruction in the Optum Healthcare Population
Brief Title: Mohs Micrographic Surgery and Reconstruction in the Optum Insurance Claims Database
Status: Withdrawn | Type: Observational
Why Stopped: The researchers were unable to answer the study question by utilizing the insurance claims database.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 832285
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Skin Cancer; Mohs Micrographic Surgery; Interpolated Flap Repair
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients from the existing Optum insurance claimed database with a confirmed diagnosis of melanoma, basal cell carcinoma, or squamous cell carcinoma who have undergone skin cancer excision surgery followed by interpolated flap repair between the years 2001-2006.

SUMMARY:
Mohs micrographic surgery (MMS) followed by skin reconstruction has been widely accepted for treatment of many skin cancers. To further characterize the trends in MMS and reconstruction for skin cancer, a retrospective analysis will be performed using the Optum© Clinformatics® DataMart de-identified commercial claims database from 2001-2016. The findings may provide critical data for future prospective studies in skin cancer treatments.

ELIGIBILITY:
Inclusion criteria:

- All patients in the Optum© Clinformatics® database who have an ICD9 or ICD10 code for skin cancer and a corresponding CPT code specific for interpolated flap reconstruction

Exclusion criteria:

- All patients for whom cost data is missing in the Optum© Clinformatics® DataMart

Ages: 1 Year to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population was conveniently sampled from the compilation of de-identified claims in the Optum© Clinformatics® database using ICD9 and ICD10 codes specific for skin cancer and linking them to specific CPT codes for interpolated flap repair, a reconstructive skin surgery. The investigator's population is composed of >7,000 patients across the United States who received a skin cancer diagnosis and this procedure between 2001 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Primary cost | Claims from 2001-2016 will be analyzed
  How does interpolation flap procedure cost differ across settings

SECONDARY OUTCOMES:
Predictors of inpatient vs. outpatient procedure | Claims from 2001-2016 will be analzyed
  How does medical specialty or geographical location predict where the procedure is performed

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Etzkorn, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No